CLINICAL TRIAL: NCT05245396
Title: A Phase I, Single-site, Open-label, Partially Randomized Study to Evaluate the Relative Bioavailability and Pharmacokinetics of Evobrutinib Following Administration of Different Formulations in Healthy Participants
Brief Title: Study Comparing Pharmacokinetics of Different Formulations of Evobrutinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS200527_0091; 2021-005056-11 (EudraCT Number)
Record Dates: First submitted 2022-01-24; First posted 2022-02-18 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: Bruton's tyrosine kinase; delayed release; multiparticulate

STUDY DESIGN:
Intervention Model Description: Part A, B and C, periods 1 to 3 will be an incomplete cross-over; Part A, B and C, periods 4 and 5 are sequential. Part D, periods 1 and 2 will be 2-sequence cross-over design with 2 treatment sequences; Part D, period 3 is optional.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part A: Evobrutinib: Treatment Sequence 1 (Experimental): Participants will receive single oral dose of modified release evobrutinib tablet-1 (MR-T1) on Day 1 in treatment period 1, followed by single oral dose of modified release tablet-2 (MR-T2) on Day 1 in treatment period 2, followed by two single oral doses of immediate release (IR) oral tablet [Ref (TF2)] on Day 1 in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or multiparticulate system capsules (MUPS-C) formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MR-T1; Drug: Evobrutinib MR-T2
- Part A: Evobrutinib: Treatment Sequence 2 (Experimental): Participants will receive single oral dose of MR-T2 on Day 1 in treatment period 1, followed by two single oral doses of Ref (TF2) on Day 1 in treatment period 2, followed by single oral dose of MR-T1 on Day 1 in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MR-T1; Drug: Evobrutinib MR-T2
- Part A: Evobrutinib: Treatment Sequence 3 (Experimental): Participants will receive two single oral doses of Ref (TF2) on Day 1 in treatment period 1, followed by single oral dose of MR-T1 on Day 1 in treatment period 2, followed by single oral dose of MR-T2 on Day 1 in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MR-T1; Drug: Evobrutinib MR-T2
- Part A: Evobrutinib: Treatment Sequence 4 (Experimental): Participants will receive single oral dose of modified release evobrutinib tablet-3 (MR-T3) on Day 1 in treatment period 1, followed by single oral dose of modified release tablet-4 (MR-T4) on Day 1 in treatment period 2, followed by two single oral doses of immediate release (IR) oral tablet [Ref (TF2)] on Day 1 in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or multiparticulate system capsules (MUPS-C) formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MR-T3; Drug: Evobrutinib MR-T4
- Part A: Evobrutinib: Treatment Sequence 5 (Experimental): Participants will receive single oral dose of MR-T4 on Day 1 in treatment period 1, followed by two single oral doses of Ref (TF2) on Day 1 in treatment period 2, followed by single oral dose of MR-T3 on Day 1 in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MR-T3; Drug: Evobrutinib MR-T4
- Part A: Evobrutinib: Treatment Sequence 6 (Experimental): Participants will receive two single oral doses of Ref (TF2) on Day 1 in treatment period 1, followed by single oral dose of MR-T3 on Day 1 in treatment period 2, followed by single oral dose of MR-T4 on Day 1 in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MR-T3; Drug: Evobrutinib MR-T4
- Part B: Evobrutinib: Treatment Sequence 1 (Experimental): Participants will receive single oral dose of MUPS-C1 evobrutinib on Day 1 in treatment period 1, followed by single oral dose of MUPS-C2 on Day 1 in treatment period 2, followed by two single oral doses of Ref (TF2) on Day 1 of in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MUPS-C1; Drug: Evobrutinib MUPS-C2
- Part B: Evobrutinib: Treatment Sequence 2 (Experimental): Participants will receive single oral dose of MUPS-C2 evobrutinib on Day 1 in treatment period 1, followed by two single oral doses of Ref (TF2) on Day 1 in treatment period 2, followed by single oral dose of MUPS-C2 on Day 1 of in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MUPS-C1; Drug: Evobrutinib MUPS-C2
- Part B: Evobrutinib: Treatment Sequence 3 (Experimental): Participants will receive two single oral doses of Ref (TF2) evobrutinib on Day 1 in treatment period 1, followed by single oral dose of MUPS-C1 on Day 1 in treatment period 2, followed by single oral dose of MUPS-C2 on Day 1 of in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MUPS-C1; Drug: Evobrutinib MUPS-C2
- Part C: Evobrutinib: Treatment Sequence 4 (Experimental): Participants will receive single oral dose of MUPS-C3 evobrutinib on Day 1 in treatment period 1, followed by single oral dose of MUPS-C4 on Day 1 in treatment period 2, followed by two single oral doses of Ref (TF2) on Day 1 of in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MUPS-C3; Drug: Evobrutinib MUPS-C4
- Part C: Evobrutinib: Treatment Sequence 5 (Experimental): Participants will receive single oral dose of MUPS-C4 evobrutinib on Day 1 in treatment period 1, followed by two single oral doses of Ref (TF2) on Day 1 in treatment period 2, followed by single oral dose of MUPS-C3 on Day 1 of in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MUPS-C3; Drug: Evobrutinib MUPS-C4
- Part C: Evobrutinib: Treatment Sequence 6 (Experimental): Participants will receive two single oral doses of Ref (TF2) evobrutinib on Day 1 in treatment period 1, followed by single oral dose of MUPS-C3 on Day 1 in treatment period 2, followed by single oral dose of MUPS-C4 on Day 1 of in treatment period 3, followed by 2 sequential periods 4 and 5. The best MR-T and /or MUPS-C formulation from period 1, 2, and 3 will be tested with additional optimization to choose the best overall formulation in treatment period 4. The best overall formulation from Period 4 may be further tested in treatment period 5 under fed or fasted conditions. There will be 72 hours washout period between Periods 1 to 3 and 28 days between Period 3 and 4 and Period 4 and 5.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MUPS-C3; Drug: Evobrutinib MUPS-C4
- Part D: Evobrutinib: Treatment Sequence 1 (Experimental): Participants will receive single oral dose of MR-T adapted on Day 1 of treatment period 1, followed by two single oral doses of Ref (TF2) on Day 1 in treatment period 2, followed by 1 sequential period 3. There will be 72 hours washout period between Periods 1 and 2 and 28 days between Period 2 and 3.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MR-T1; Drug: Evobrutinib MR-T adapated
- Part D: Evobrutinib: Treatment Sequence 2 (Experimental): Participants will receive two single oral doses of Ref (TF2) on Day 1 of treatment period 1, followed by single oral dose of MR-T adapted on Day 1 in treatment period 2, followed by 1 sequential period 3. There will be 72 hours washout period between Periods 1 and 2 and 28 days between Period 2 and 3.
  Interventions: Drug: Ref (TF2); Drug: Evobrutinib MR-T1; Drug: Evobrutinib MR-T adapated

INTERVENTIONS:
Drug: Ref (TF2) — Participants will receive 2 single oral doses of Ref (TF2) on Day 1 in treatment period 1, 2, or 3 of Part A, B, C and D.
  Other Names: M2951
Drug: Evobrutinib MR-T1 — Participants will receive single oral dose of MR-T1 on Day 1 in treatment period 1, 2, and 3 of Part A.
  Other Names: M2951
  Arms: Part A: Evobrutinib: Treatment Sequence 1; Part A: Evobrutinib: Treatment Sequence 2; Part A: Evobrutinib: Treatment Sequence 3; Part D: Evobrutinib: Treatment Sequence 1; Part D: Evobrutinib: Treatment Sequence 2
Drug: Evobrutinib MR-T2 — Participants will receive single oral dose of MR-T2 on Day 1 in treatment period 1, 2, and 3 of Part A.
  Other Names: M2951
  Arms: Part A: Evobrutinib: Treatment Sequence 1; Part A: Evobrutinib: Treatment Sequence 2; Part A: Evobrutinib: Treatment Sequence 3
Drug: Evobrutinib MR-T3 — Participants will receive single oral dose of MR-T3 on Day 1 in treatment period 1, 2, and 3 of Part A.
  Other Names: M2951
  Arms: Part A: Evobrutinib: Treatment Sequence 4; Part A: Evobrutinib: Treatment Sequence 5; Part A: Evobrutinib: Treatment Sequence 6
Drug: Evobrutinib MR-T4 — Participants will receive single oral dose of MR-T4 on Day 1 in treatment period 1, 2, and 3 of Part A.
  Other Names: M2951
  Arms: Part A: Evobrutinib: Treatment Sequence 4; Part A: Evobrutinib: Treatment Sequence 5; Part A: Evobrutinib: Treatment Sequence 6
Drug: Evobrutinib MUPS-C1 — Participants will receive single oral dose of MUPS-C1 on Day 1 in treatment period 1, 2, and 3 of Part B.
  Other Names: M2951
  Arms: Part B: Evobrutinib: Treatment Sequence 1; Part B: Evobrutinib: Treatment Sequence 2; Part B: Evobrutinib: Treatment Sequence 3
Drug: Evobrutinib MUPS-C2 — Participants will receive single oral dose of MUPS-C2 on Day 1 in treatment period 1, 2, and 3 of Part B.
  Other Names: M2951
  Arms: Part B: Evobrutinib: Treatment Sequence 1; Part B: Evobrutinib: Treatment Sequence 2; Part B: Evobrutinib: Treatment Sequence 3
Drug: Evobrutinib MUPS-C3 — Participants will receive single oral dose of MUPS-C3 on Day 1 in treatment period 1, 2, and 3 of Part C.
  Other Names: M2951
  Arms: Part C: Evobrutinib: Treatment Sequence 4; Part C: Evobrutinib: Treatment Sequence 5; Part C: Evobrutinib: Treatment Sequence 6
Drug: Evobrutinib MUPS-C4 — Participants will receive single oral dose of MUPS-C4 on Day 1 in treatment period 1, 2, and 3 of Part C.
  Other Names: M2951
  Arms: Part C: Evobrutinib: Treatment Sequence 4; Part C: Evobrutinib: Treatment Sequence 5; Part C: Evobrutinib: Treatment Sequence 6
Drug: Evobrutinib MR-T adapated — Participants will receive single oral dose of MR-T adapted on Day 1 in treatment period 1, 2, and 3 of Part D.
  Other Names: M2951
  Arms: Part D: Evobrutinib: Treatment Sequence 1; Part D: Evobrutinib: Treatment Sequence 2

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK), pharmacodynamic (PD), and safety and tolerability of evobrutinib after oral administration of immediate release (IR) and modified release (MR) formulations in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as determined by medical evaluation, including comprehensive clinical assessment (detailed medical history and a complete physical examination), ECG, and laboratory investigations (hematology and biochemistry)
* Participants have a body weight within 50.0 to 100.0 kilogram (kg) and body mass index (BMI) within the range 19 to 32 kilogram per meter square (kg/m^2) (inclusive)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with history or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, metabolic, hematological, lymphatic, neurological (including epilepsy), cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, as determined by medical evaluation
* Participants with history of any malignancy
* Administration of live vaccines or live-attenuated virus vaccines within 3 months prior to Screening. Administration of other types of vaccines (e.g. SARS-CoV-2 vaccines) is allowed until 2 weeks before the admission to the CRU
* Medical history and physical examination results that include any ongoing clinically relevant findings as judged by the Investigator
* Moderate or strong inhibitors or inducers of CYP3A4/5 or Pgp within 4 weeks prior to the first administration of study intervention
* Other protocol-defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability Based on Area Under the Plasma Concentration Curve From Time Zero to 24 Hours Post Dose [Frel(AUC0-24)] of Evobrutinib Modified-Release Formulation Compared to Immediate-Release Evobrutinib Reference Formulation | Pre-dose up to 72 hours post-dose on Day 4
Relative Bioavailability Based on Area Under the Plasma Concentration Curve From Time Zero to Infinity [Frel(AUC0-inf)] of Evobrutinib Modified-Release Formulation Compared to Immediate-Release Evobrutinib Reference Formulation | Pre-dose up to 72 hours post-dose on Day 4

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), Abnormal Laboratory Test Results, Abnormal Vital Signs and Abnormal Electrocardiogram (ECG) Measurements | Up to Day 123
Pharmacokinetic Plasma Concentration of Evobrutinib Formulations | Pre-dose up to 72 hours post-dose on Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Quotient Clinical Ltd, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0091
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html